CLINICAL TRIAL: NCT04282694
Title: PRogetto Salute Parma: PRevenzione Primaria e Secondaria Del Danno da Fumo
Brief Title: PRogetto Salute Parma
Acronym: PSP
Status: Terminated | Type: Observational
Why Stopped: The worldwide surge of SARS-CoV-2 started during the first week of the study. The Investigators attempted to re-organize the project with a new agenda, but the time frame from the funding Organization did not comply with the study needs.
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Unità Sanitaria Locale di Parma (Other)
Responsible Party: Sponsor
Other Study IDs: 837/2019/OSS/UNIPR
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2020-02

CONDITIONS: Smoking; Smoking Habit; Smoking, Tobacco; Smoking, Cigarette; Smoking Cessation; Lung Cancer
MeSH Terms: conditions — Smoking; Tobacco Smoking; Cigarette Smoking; Smoking Cessation; Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- High risk (former) smokers: Subjects at high risk of lung cancer screened by the medical team of the AOUPR or by GPs to join the prevention program.
  Inclusion criteria
  * Age between 50 and 75 years
  * Equivalent tobacco intoxication of ≥ 15 cigarettes per day for ≥25 years or ≥ 10 cigarettes per day for ≥30 years
  * Status of current smoker or ex-smoker for <10 years.
  Exclusion criteria
  • Personal history of cancer within the prior 5 years
  Interventions: Diagnostic Test: Low-dose computed tomography (LDCT)

INTERVENTIONS:
Diagnostic Test: Low-dose computed tomography (LDCT) — Early detection of lung cancer by LDCT and smoking cessation counselling
  Other Names: Smoking cessation

SUMMARY:
This project from the University Hospital of Parma (AOUPR) aims to verify the feasibility of a prevention program in our district, relying on advanced technological resources and highly experienced team in lung cancer early diagnosis, in order to identify useful elements towards the applicability of such a prevention program on a large scale (regional, national).

Uncontrolled, monocentric experimental study with dynamic enrollment and prospective data collection, aimed at implementing a prevention program based on scientific evidence. This study is set to verify the applicability and feasibility of a lung cancer prevention program in a real context, including a preliminary evaluation at the smoking cessation clinic and a LDCT assessment with subsequent LDCT follow-up for participants who show indeterminate findings at the first LDCT (LDCT baseline) exam.

The main objective of the study is to verify the feasibility of a lung cancer prevention program according to internationally validated scientific methods.

Secondary objectives:

1. To evaluate the use of local smoking cessation clinics and their effects in terms of smoking cessation (primary prevention)
2. To evaluate the outcomes of the program in terms of number of patients with early (presymptomatic) lung cancer treated with minimally invasive surgery (secondary prevention)
3. To evaluate the number of false positives and their diagnostic work-up (PET-CT, CT-guided biopsy, bronchoscopy)

Primary endpoint:

- Percentage of enrolled subjects to whom the program was offered within 60 days from the date of enrolment and percentage of those who stop smoking for at least 12 months

Secondary endpoints:

* To describe the organizational model, human resources employed, difficulties encountered and elements that have favoured its realization
* To measure the variation in smoking habits in enrolled smokers
* To describe the effect of annual LDCT on lung cancer diagnosis rates, considering size, shape, histology and site
* To measure the consequent demand for further diagnostic investigations and treatment
* To measure the number of false positives

Subjects at high risk of lung cancer screened by the medical team of the AOUPR or by GPs to join the prevention program.

Inclusion criteria

* Age between 50 and 75 years
* Equivalent tobacco intoxication of ≥ 15 cigarettes per day for ≥25 years or ≥ 10 cigarettes per day for ≥30 years
* Status of current smoker or ex-smoker for <10 years.

Exclusion criteria

• Personal history of cancer within the prior 5 years

We expect to recruit around 500 people in 1 year. This sample size is considered adequate based on the available resources, both human and economic.

After closing and adjusting the database and before data analysis, a document called Statistical Analysis Plan (SAP) will be drawn up. It will consist of the following paragraphs:

* Statistical methods planned in the study protocol;
* Size of the sample;
* Management of missing data;
* Evaluation of the endpoints;
* Statistical models that will be applied in the analysis. The socio-demographic characteristics of the enrolled subjects, the adopted organizational methods and the effects of the prevention program (endpoints) will be analyzed and described using tables and figures.

The project "PRogetto Salute Parma: Primary and secondary prevention of smoking-related lung cancer" will be started once approved by the institutional Ethics Committee and authorized by the General Manager. The study is expected to be carried out over 2 years (from the inclusion of the first subject), with an expected period of 1 year for the enrolment and 1 further year for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Equivalent tobacco intoxication of ≥ 15 cigarettes per day for ≥25 years or ≥ 10 cigarettes per day for ≥30 years
* Status of current smoker or ex-smoker for <10 years.

Exclusion Criteria:

* Personal history of cancer within the prior 5 years

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We expect to recruit around 500 people in 1 year. This sample size is considered adequate based on the available resources, both human and economic.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Adherence | 12 months
  Percentage of enrolled subjects to whom the program was offered within 60 days from the date of enrolment and percentage of those who stop smoking for at least 12 months

SECONDARY OUTCOMES:
Organization model | 18 months
  To describe the organizational model, human resources employed, difficulties encountered and elements that have favoured its realization
Smoking cessation | 24 months
  To measure the variation in smoking habits in enrolled smokers.
Secondary prevention of lung cancer | 24 mesi
  To describe the effect of annual LDCT on lung cancer diagnosis rates, considering size, shape, histology and site.
Work up burden | 24 months
  To measure the demand for further diagnostic investigations and treatment generated by LDCT.
False positives | 24 months
  To measure the number of false positives generated by LDCT

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Sverzellati, MD, PhD, Principal Investigator — University of Parma
Locations (1):
- University of Parma, Parma, Italy